CLINICAL TRIAL: NCT04614142
Title: Single Patient Protocol for Donor HCV-positive to Recipient HCV-negative Kidney Transplant in a Patient at Risk for Loss of Dialysis Access
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Single patient the protocol was written for consented to another study.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology and Liver Center, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020P003265
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease; Chronic Hepatitis c
Keywords: kidney transplantation; hepatitis C; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Glecaprevir/pibrentasvir for HCV+ kidney transplant recipient (Experimental): Glecaprevir (100mg) / pibrentasvir (40mg) (fixed dose combination) treatment for Hepatitis C virus (HCV)-naive recipients who receive a kidney transplant from a deceased, HCV-infected donor.
  Subject will receive first dose on day 3 (+/- 2 days) post-kideny transplantation and continue daily for 8 weeks.
  Interventions: Drug: Glecaprevir / Pibrentasvir Oral Tablet [Mavyret]

INTERVENTIONS:
Drug: Glecaprevir / Pibrentasvir Oral Tablet [Mavyret] — The subject will begin an 8 week course of therapy with glecaprevir (100mg) / pibrentasvir (40mg) starting on day 3 (+/- 2 days) post-kidney transplantation from a hepatitis C positive donor.

SUMMARY:
This is a single patient, single center study evaluating if administration of pan-genotypic DAA therapy on day 3 (+/- 2 days) post-kidney transplant prevents the transmission of hepatitis C virus infection from an HCV-positive donor kidney to an HCV-negative recipient.

DETAILED DESCRIPTION:
The patient selected for this study previously received a kidney transplant under protocol 2016P002051. Unfortunately, she experienced primary graft nonfunction due to a renal vein thrombus and acute thrombotic microangiopathy and the transplanted HCV+ kidney was removed. She continued glecaprevir and pibrentasvir for the full course (8 weeks of treatment) and was cured of HCV. However, she continues on dialysis requiring ongoing, albeit low dose, immunosuppression after her failed transplant. This causes increased risk of infection and other dialysis-related morbidity. Futhermore, she is at risk of access loss due to multiple failed fistula attempts and prior dialysis catheter line thrombosis. Of note, she also failed a trial of peritoneal dialysis due to development of a large pleural effusion (a known treatment-limiting complication of peritoneal dialysis). Thus, this young patient, is at risk of losing dialysis access which could lead to death. The MGH transplant team has now decided that she could be retransplanted with alterations in peri-transplant anticoagulation and immunosuppression (eculizumab) that they are confident should decrease her risk of peri-transplant thrombosis and recurrent TMA. Thus, we desire to expedite her access to re-transplant. Through this protocol, this recipient will be given the opportunity to accept a kidney that is HCV antibody positive and nucleic acid test (NAT) negative or HCV NAT positive and will be treated with oral glecaprevir (300mg)/pibrentasvir (120mg) (G/P, MavyretTM) on day 3 (+/- 2 days) post-kidney transplant to prevent the transmission of HCV infection at the time of transplant. Our goal is to provide access to kidney transplantation as soon as possible, with a donor of any genotype of infection, with elimination of the potential HCV infection by therapy used on day 3 (+/- 2 days) in the case of HCV NAT+ transplant and surveillance and reactive therapy in the case of HCV antibody positive NAT- transplant.

ELIGIBILITY:
Donor Inclusion Criteria:

* Detectable HCV Antibody Positivity
* KDPI score is less than ≤ 0.650
* Traditional Donor Selection Criteria Met - acceptable for transplantation per usual evaluation at MGH

Donor exclusion criteria

* Donor has been known to have previously received and failed HCV treatment with a direct-acting antiviral agent
* Confirmed HIV
* Confirmed HBV positive (surface antigen or HBV DNA positive)
* Kidney anatomical damage or significant pathology noted during recovery
* Significant liver disease or signs of liver decompensation (splenomegaly, ascites) noted during recovery (advanced fibrosis or cirrhosis)
* Any standard contra-indication to donation noted in donor (significant malignancy, unusual infection)

Recipient Inclusion/Exclusion Criteria

* Previously enrolled in IRB 2016P002051 and experienced primary graft nonfunction due to renal vein thrombosis and acute thrombotic microangiopathy
* Willing and able to sign informed consent

Ages: 34 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-selected subject is female
Enrollment: 0 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Hepatitis C viral load (RNA) | 20 weeks post-transplant (12-weeks post-treatment)
  Negative hepatitis C viral load (RNA) tested using PCR at 12 weeks post-treatment (SVR12)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside of the research team.

REFERENCES:
- [Background] Goldberg DS, Abt PL, Blumberg EA, Van Deerlin VM, Levine M, Reddy KR, Bloom RD, Nazarian SM, Sawinski D, Porrett P, Naji A, Hasz R, Suplee L, Trofe-Clark J, Sicilia A, McCauley M, Farooqi M, Gentile C, Smith J, Reese PP. Trial of Transplantation of HCV-Infected Kidneys into Uninfected Recipients. N Engl J Med. 2017 Jun 15;376(24):2394-2395. doi: 10.1056/NEJMc1705221. Epub 2017 Apr 30. No abstract available. PMID 28459186
- [Background] Reau N, Kwo PY, Rhee S, Brown RS Jr, Agarwal K, Angus P, Gane E, Kao JH, Mantry PS, Mutimer D, Reddy KR, Tran TT, Hu YB, Gulati A, Krishnan P, Dumas EO, Porcalla A, Shulman NS, Liu W, Samanta S, Trinh R, Forns X. Glecaprevir/Pibrentasvir Treatment in Liver or Kidney Transplant Patients With Hepatitis C Virus Infection. Hepatology. 2018 Oct;68(4):1298-1307. doi: 10.1002/hep.30046. Epub 2018 Jul 25. PMID 29672891
- [Background] Durand CM, Bowring MG, Brown DM, Chattergoon MA, Massaccesi G, Bair N, Wesson R, Reyad A, Naqvi FF, Ostrander D, Sugarman J, Segev DL, Sulkowski M, Desai NM. Direct-Acting Antiviral Prophylaxis in Kidney Transplantation From Hepatitis C Virus-Infected Donors to Noninfected Recipients: An Open-Label Nonrandomized Trial. Ann Intern Med. 2018 Apr 17;168(8):533-540. doi: 10.7326/M17-2871. Epub 2018 Mar 6. PMID 29507971
- [Background] Sise ME, Goldberg DS, Kort JJ, Schaubel DE, Alloway RR, Durand CM, Fontana RJ, Brown RS Jr, Friedewald JJ, Prenner S, Landis JR, Fernando M, Phillips CC, Woodle ES, Rike-Shields A, Sherman KE, Elias N, Williams WW, Gustafson JL, Desai NM, Barnaba B, Norman SP, Doshi M, Sultan ST, Aull MJ, Levitsky J, Belshe DS, Chung RT, Reese PP. Multicenter Study to Transplant Hepatitis C-Infected Kidneys (MYTHIC): An Open-Label Study of Combined Glecaprevir and Pibrentasvir to Treat Recipients of Transplanted Kidneys from Deceased Donors with Hepatitis C Virus Infection. J Am Soc Nephrol. 2020 Nov;31(11):2678-2687. doi: 10.1681/ASN.2020050686. Epub 2020 Aug 25. PMID 32843477